CLINICAL TRIAL: NCT05321641
Title: Evaluation Of A Mobile Messaging Service (Text And / Or Graphic) In Improving Adherence With Ensured Supply Of Anti-Seizure Medications In People With Epilepsy In Kilifi And Nairobi, Kenya
Brief Title: Evaluation Of A Mobile Messaging Service In Improving Adherence Of Anti-Seizure Medications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: KEMRI-Wellcome Trust Collaborative Research Program (Other)
Collaborators: University of Oxford (Other); African Population and Health Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: KEMRI 4368
Record Dates: First submitted 2022-03-07; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Epilepsy; Treatment Adherence
MeSH Terms: conditions — Epilepsy; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: We plan to randomize 1200 people with epilepsy at each site, from a defined area in Kilifi and Nairobi County, Kenya. They will be divided into four groups of 300 each, to receive either text SMS, graphic SMS, both text and graphic or SMS on public health promotion not related to epilepsy e.g. use of bednets (for comparison).
Who Masked: Investigator, Outcomes Assessor
Masking Description: The participants can tell if they are receiving adherence messages or general public health messages. The clinicians will interact with participants and may therefore get to know what kind of messages they receive. However, the investigators, who will conduct the analysis and the assessors will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Text SMS (Experimental): Adherence messages presented in both text form.
  Interventions: Behavioral: Mobile phone message reminders.
- Graphic SMS (Experimental): Adherence messages presented in graphic form.
  Interventions: Behavioral: Mobile phone message reminders.
- Both text and graphic (Experimental): Adherence messages presented in both text and graphic form.
  Interventions: Behavioral: Mobile phone message reminders.
- Control (Placebo Comparator): Messages on public health promotion not related to epilepsy
  Interventions: Behavioral: Mobile phone message reminders.

INTERVENTIONS:
Behavioral: Mobile phone message reminders. — Utilising mobile messaging service to send reminders to people with epilepsy to take antiseizure medications and sending reminders to primary health facilities to restock anti-seizure medications.

SUMMARY:
This will be a behavioural intervention with no investigational medicinal product.

The intervention will be a mobile messaging service that sends short messaging service (SMS) as texts or graphics to people with epilepsy to remind them to take their medication and to refill their prescription and educational messages to share important messages tackling stigma and tips to improve quality of life.

The investigators will also engage peripheral health facilities where people with epilepsy (PWE) participating in the study go for ASM refills, in collaboration with the respective county departments of health, to maintain adequate supply of anti-seizure medications through:

i. ongoing capacity building studies in Kilifi such as the mental health Gap Action Programme-Intervention Guide (mhGAP-IG) training which is empowering primary healthcare providers at peripheral health facilities to identify and manage epilepsy and other mental health disorders. ii. supporting healthcare providers at peripheral facilities through in person visits, if the COVID-19 situation, permits or by telephone or standard message reminders to restock their ASM supply.

The participants in the no-intervention group will receive "placebo" health messages not related to epilepsy such as use of bednets. The SMS reminders will be sent at a frequency that will be agreed upon during pre-study engagements with potential participants, whether daily, weekly, or monthly. The participants will be able to respond to these texts to report on their health status and any adverse events.

To evaluate whether SMS reminders improve adherence, we will use: i. Self-reporting adherence scales- the Morisky Medication Adherence Scale (MMAS-8) ii. Measurement of ASM plasma levels at 12 months from baseline.

DETAILED DESCRIPTION:
Improved outcomes for epilepsy treatment depend on a continuous supply and daily adherence to anti-seizure medications (ASMs). In Kilifi County, the treatment gap which includes both the diagnostic and adherence gap, is greater than 70% and investigators have found interruption of supply of ASMs to peripheral clinics, distance from clinic and lack of availability of ASMs, to be barriers to adherence. In Nairobi County, factors such as environment hazards, lack of social amenities and correlates of poverty are preponderant in slums, but the prevalence of epilepsy has not been studied in such settings and consequently, the adherence gap remains unknown. Innovative mobile Health (mHealth) strategies including messages delivered by mobile phones have been used to ensure an adequate supply of drugs in health centres, and daily mobile messages have improved adherence to medication in Human Immunodeficiency Virus (HIV) programs, for example. Text messaging requires that the patient has access to a mobile phone and can understand the text message. Multimedia messaging, such as simple pictures, may improve understanding of the necessity to take medication, particularly in people who are illiterate, and we will explore this as an avenue to improve uptake.

The investigators plan to randomize 1200 people with epilepsy at each site, from a defined area in Kilifi and Nairobi County, Kenya. They will be divided into four groups of 300 each, to receive either text SMS, graphic SMS, both text and graphic or SMS on public health promotion not related to epilepsy e.g. use of bednets (for comparison). The investigators aim is to i) describe the perceptions and perspectives of people with epilepsy and their caregivers on the use of text and graphic SMS reminders to improve adherence to ASMs, ii) compare the effectiveness of text versus graphic messaging service in improving adherence in people with epilepsy and to engage the County Departments of Health through current ongoing training and capacity building studies to maintain supply of ASMs in peripheral clinics iii) identify the factors associated with improvement in adherence, improved QoL and reduction in stigma among people with epilepsy and family members and iv) conduct cost-effectiveness assessment for the roll out of the intervention. Besides medication-related messages, there will be other messages, from previous community-based feedback, selected to address stigmatization and improve quality of life. Blood-level monitoring and adherence questionnaires at baseline and during subsequent follow up visits will be used to assess as measures of medication adherence. If found useful, this intervention may be applicable for self-managing other chronic conditions in under-resourced settings.

ELIGIBILITY:
Inclusion Criteria:

* Children or adults with a diagnosis of epilepsy ascertained by a clinician at the epilepsy clinic
* Taking anti-seizure medications at the time of the study
* Living within an area defined as the Kilifi Health Demographic Surveillance System, or the Nairobi Urban Health and Demographic Surveillance System at the time of the study or attending the epilepsy clinic in Kilifi or a KAWE-led clinic in Nairobi
* Able to give written informed consent or assent in addition to parental consent (if aged between 13 and 17 years old) to participate in the study either by themselves or in the presence of an independent witness

Exclusion Criteria:

* Have intellectual disability
* Do not have access to basic mobile phones
* Are currently enrolled in ongoing interventions aimed at improving their health care

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Adherence to anti-seizure medications | 12 months since baseline.
  This will be measured through self-reports scales (eg the Morisky Medication Adherence Scale (MMAS-8)), checking record logs for correct intake of drugs and refill rates- validated by optimal and detectable levels in blood.

SECONDARY OUTCOMES:
Changes in seizure frequency, from many seizures to fewer seizures. | 12 months since baseline.
  These will be assessed by trained clinicians at the epilepsy clinics, through routine clinical examination.
Changes in stigma scores and quality of life scores, from higher scores to less scores for stigma and from lower scores to higher scores for quality of life. | 12 months since baseline.
  These will be assessed with standardized and locally adapted scales (assessed with the Kilifi Epilepsy Stigma Scale and World Health Organization Quality of Life Scale (WHOQOL-BREF), respectively).

OTHER OUTCOMES:
Pharmacovigilance for unwanted drug-related adverse events as reported by participants and confirmed using standardized questionnaire. | 12 months since baseline.
  Many patients will be on old generation anti-seizure medications which have undesirable effects, so systematic monitoring of adverse events using Common Toxicity Criteria for Adverse Events (CTCAE) is important.

CONTACTS AND LOCATIONS:
Overall Officials: Charles R Newton, MD, Study Director — KEMRI-Wellcome Trust Collaborative Research Program; Symon M Kariuki, DPhil, Principal Investigator — KEMRI-Wellcome Trust Collaborative Research Program; Arjune Sen, PhD, Principal Investigator — University of Oxford
Locations (1):
- KEMRI Wellcome Trust Research Programme, Kilifi, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Individual-level anonymized data will be shared with the Sponsor. Summary-level statistical analyses will be shared with wider stakeholder engagement and the medical community.
  Information collected or generated during this study may be anonymised for use to support new research on epilepsy. Any future research using information from this study must first be approved by a local or national expert committee to make sure that the interests of participants and their communities are protected. Data will be managed by the data governance committee of KEMRI CGMRC.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From 2-5 years after the study completion.
Access Criteria: Approved proposal and analysis plan and permission to access the data from the data governance committee.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT05321641/Prot_SAP_000.pdf